CLINICAL TRIAL: NCT03846882
Title: The Value of PET / MRI for the Assessment of Lymph Node Metastasis and Other Prognostic Factors in Patients With Rectal Cancer
Brief Title: FDG - PET / MRI in Patients With Rectal Cancer
Acronym: RECTOPET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Katrine Riklund, MD; PhD, Clinical Professor, Consultant, Principal Investigator, Region Västerbotten
Other Study IDs: 2015-417-31
Record Dates: First submitted 2018-07-06; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Rectal Cancer; Lymph Node Metastases
Keywords: PET/MR; PET/CT; FDG; Staging
MeSH Terms: conditions — Rectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The combination of FDG-PET/CT and MRI at staging of rectal cancer in diagnosis is currently very little studied. The investigator have a unique opportunity to study this. Hypothetically, with PET/MR as one hybrid imaging method, alternatively as an additional method, it could increase the accuracy of rectal cancer of moderate and high risk type, especially at primary N-staging, but also in assessing other important prognostic factors such as T-staging, peritoneal involvement, metastasis to lateral lymph nodes, EMVI and MRF involvement. The same reasoning applies to the assessment of tumor regression after CRT.

In the study, PET/MR is compared with PET/CT, diagnostic CT and MRI to evaluate the additional value of the hybrid imaging PET/MRI. The investigator also plan to evaluate how immunological, proliferative and prognostic biomarkers in blood and tumor tissue correlate with the radiological findings, and if the combination biomarker and radiology can provide additional prognostic information.

DETAILED DESCRIPTION:
Today, there is a variety of treatment options in diagnosed rectal cancer. The standard treatment is surgery with removal of the tumour including surrounding fat and lymph nodes in a package. Prior to surgery, the patient may be given a shorter or longer radiation treatment, the latter in combination with cytostatics, depending on staging at the time of diagnosis. Cytostatic drugs can also be given post surgery. The choice of treatment for the individual patient is based on the assessment of the imaging, ie conventional X-ray, ultrasound, computed tomography, (CT), Magnet Resonance Tomography Imaging (MRI) and Positron Emission Tomography in combination with CT (PET/CT). An accurate staging assessment is crucial for adequate treatment of rectal cancer patients to avoid over treatment, which in itself causes unnecessary suffering, or under treatment with increased risk of relapse. With today's methods, tumor size, overgrowth of other organs and spread to other organs such as liver and lung can be reasonable assessed. On the other hand, there is great uncertainty when assessing spread to lymph nodes. Better safety is also needed for other prognostically important factors such as tumor involvement of the mesorectal fasciae (MRF), i.e. the rectum surrounding the tumor, and tumor growth in venous vessels outside the intramural invasion of the intestinal wall, EMVI.

Hybrid imaging with PET combined with magnetic resonance imaging (PET/MR) is a novel method and there are currently no published studies comparing the outcome of fluoro-deoxy glucose (FDG) -PET/MR with CT, MR, PET/CT at staging of rectal cancer, both primarily and after radiation and cytostatics treatment (CRT). In this study, the investigator plan to evaluate the additional value for PET/MR in rectal cancer. Only patients to be operated are included and microscopic examination of the preparation, histopathology, will be the reference method with which survey data from the imaging methods are compared. The investigator also want to evaluate the relationship between the radiological findings and biomarkers in blood and tumor tissue to determine if there is a relationship that can provide additional prognostic information. The investigator will only include patients with intermediate and high-risk rectal cancer, as low-risk cancer is unusual with spread to lymph nodes. The study will be a prospective observation study in which all consecutive elective patients in Umeå with confirmed intermediate and high risk type rectal cancer, which give their consent, are included and examined preoperatively. Thereafter, imaging and blood and tumor tissue samples are examined and evaluated.

Primary research questions:

* Can FDG-PET/MR provide improved accuracy in assessment of local tumor proliferation, lymph node metastasis and other important prognostic factors (MRF +, EMVI) in rectal cancer compared to currently used methods magnetic resonance imaging, (MRI), PET/CT or CT?
* Can FDG-PET/MR provide an improved accuracy in assessment of tumor regression following combined cytostatics and radiotherapy in rectal cancer compared to MRI or PET/CT?
* Can FDG-PET / MR in combination with blood and tumor tissue biomarkers provide additional prognostic information for intermediate and high-risk rectal cancer?

Secondary research questions:

• How does the accumulation of FDG change in rectal cancer tissue when examined after 60 minutes vs examination after 90 minutes?

Patients will be examined with a whole body FDG-PET CT, where the CT replaces the regular diagnostic CT examination. There is also a FDG-PET/MR of the pelvic region, where the MR part replaces the regular MRI examination. For patients with locally advanced disease undergoing combined radiation and chemotherapy, a further PET/CT and PET/MR are acquired at least 4 weeks after the treatment, but before surgery. In future, patients who only need shorter radiation therapy may undergo further PET/CT and PET/MR before surgery, if time between radiation and surgery is extended as clinical routine.

PET/CT and PET/MR are done immediately after each other with only one FDG injection of 4 Mbq/kg body weight. The examinations will be reviewed and judged according to clinical routine, where all reviewers have access to all image data. An additional reading will then be done by experienced GI-radiologist and nuclear medicine physician to assess the additional value for PET/MR. The histopathological finding in the examination of the surgical preparation will be used as a reference method.

In order to facilitate the assessment and correlation between individual lymph nodes in tissue analysis and imaging data, the operation specimen will, when this is possible, be examined with MRI postoperatively before the histopathological examination is performed.

The study does not involve any extra visits in addition to clinical routine at the Department of Radiology, but gives a small increase in radiation dose, as PET/MR is done instead of MRI only and in addition to PET/CT after CRT, which is not clinical routine. According to national guidelines, PET/CT is intended for advanced rectal cancer, but for those not included in this group, there will be an increased radiation dose of PET in PET/CT. This increase of ionizing radiation is small and corresponds to approximately 2 years of background radiation.

Radiological image data (PET/MR and PET/CT) is stored in the picture archiving and communicating system (PACS) as in clinical routine. Requests and reports are stored in the Department's Radiological Information System (RIS).

The examination is subject to the same confidentiality as any routine imaging examination at the department. Image data will not be destroyed. Data is exported to external software for post processing and statistical processing. All processing in addition to clinical routine takes place in unidentified data. Only those responsible and employees in the project have access to conversion lists.

The primary objective of this study is assessment of lymph node metastases. The best method today is MR which has a sensitivity of 77% and a specificity of 71%. With an estimated 20% prevalence of lymphoma metastases, an expected sensitivity of 90%, an expected specificity of 80% and 80% statistical strength, and 95% confidence interval, 307 glands are required for sensitivity and 691 glands for specificity. As the investigator expect to identify 8 glands per patient, it means that about 39 patients is needed for the sensitivity and about 87 patients for the specificity. The investigator round up the number of patients to 100 to compensate for any failure in the follow-up.

Written information is provided to the patient and patient leaves his signature. All signed consent is given to the x-ray department where they are filed at the research department. Individuals who can not or do not want to give consent are not included. This also applies to individuals with reduced decision-making skills.

The examination is subject to the same confidentiality as any routine x-ray examination at the clinic. Evaluation of the find takes place under safe forms within a limited circle and data is kept in safe storage. If external statistical consultation is required, patient data will be unidentified.

ELIGIBILITY:
Inclusion Criteria:

* verified rectal cancer of intermediate or high risk type, scheduled for surgery (non-acute surgery)

Exclusion Criteria:

* kidney dysfunction
* any other contraindications for contrast agents or examination with MRi or FDG-PET/CT

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: With an estimated 20% prevalence of lymphoma metastases, an expected sensitivity of 90%, an expected specificity of 80% and 80% statistical strength, and 95% confidence interval, 307 glands are required for sensitivity and 691 glands for specificity. The investigator expect to identify 8 glands per patient, which means that about 39 patients for the sensitivity and about 87 patients for the specificity is needed. The investigator round up the number of patients to 100 to compensate for any failure in the follow-up.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Improved accuracy with FDG-PET/MR in assessment of local tumor proliferation, lymph node metastasis and other important prognostic factors (MRF +, EMVI) in rectal cancer compared to currently used methods MRI, PET/CT or CT? | 8years
  Sensitivity, specificity and likelihood ratios of primary and restaging FDG-PET/MR in the identification of mesorectal lymph node metastases compared to primary and restaging FDG-PET/CT, MRI and CT alone with histopathological examination as reference standard.
Improved accuracy in assessment of tumor regression following combined cytostatic and radiation treatment in rectal cancer with FDG-PET/MR compared to MRI or PET/CT? | 8years
  Sensitivity, specificity and likelihood ratios of primary and restaging FDG-PET/MR in the characterization of extramural vascular invasion and tumour deposits compared to primary and restaging FDG-PET/CT, MRI and CT alone with histopathological examination as reference standard.
Can FDG-PET / MR in combination with blood and tumor tissue biomarkers provide additional prognostic information for intermediate and high-risk rectal cancer? | 8years
  Correlation between metabolic tumor regression grading with restaging FDG-PET/MR performed after neoadjuvant chemoradiation compared to restaging FDG-PET/CT, MRI and CT alone with histopathological tumour regression grading according to TNM as reference standard.

SECONDARY OUTCOMES:
How does the accumulation of FDG change in rectal cancer tissue when examined after 60 minutes vs examination after 90 minutes? | 3years
  Correlation between Standard uptake value (SUV) mean, SUV max and total glycolytic content in rectal cancer at 60 and 90 minutes after FDG Injection in the primary tumour and lymph node metastases in the primary examinations and at restaging compared to blood and tumor tissue biomarkers and two and five-year clinical follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Riklund, MD, PhD, Principal Investigator — Department of Radiation Sciences, Diagnostic Radiology, Umeå university, Sweden
Locations (1):
- Department of Radology, Umeå, Sweden

REFERENCES:
- [Derived] Rutegard MK, Batsman M, Blomqvist L, Rutegard M, Axelsson J, Ljuslinder I, Rutegard J, Palmqvist R, Brannstrom F, Brynolfsson P, Riklund K. Rectal cancer: a methodological approach to matching PET/MRI to histopathology. Cancer Imaging. 2020 Oct 31;20(1):80. doi: 10.1186/s40644-020-00347-6. PMID 33129352
- [Derived] Rutegard MK, Batsman M, Axelsson J, Brynolfsson P, Brannstrom F, Rutegard J, Ljuslinder I, Blomqvist L, Palmqvist R, Rutegard M, Riklund K. PET/MRI and PET/CT hybrid imaging of rectal cancer - description and initial observations from the RECTOPET (REctal Cancer trial on PET/MRI/CT) study. Cancer Imaging. 2019 Jul 23;19(1):52. doi: 10.1186/s40644-019-0237-1. PMID 31337428